CLINICAL TRIAL: NCT03989375
Title: The Effect of Transcutaneous Electrical Stimulation of the Vagus Nerve on Reduction of Postoperative Cognitive Dysfunction in Elderly Patients After Hip or Knee Arthroplasty
Brief Title: Transcutaneous Electrical Stimulation of the Vagus Nerve
Acronym: TESVNR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, diansan su, Professer, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: diansansu2018013
Record Dates: First submitted 2019-06-16; First posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Cognitive Dysfunction
Keywords: postoperative Cognitive Dysfunction; hip- and knee arthroplasty; transcutaneous vagus nerve stimulation
MeSH Terms: conditions — Cognitive Dysfunction; Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Experimental)
  Interventions: Device: transcutaneous vagus nerve electric stimulator
- control group (No Intervention)

INTERVENTIONS:
Device: transcutaneous vagus nerve electric stimulator — The stimulator that can be attached to ears of the patient.We suppose that this device can reduce the incidence of perioperative neurocognitive disorders(PND)
  Arms: experiment group

SUMMARY:
This study evaluate the cognitive functions of patient after hip or kneel replacement.Half of the patient will receive transcutaneous vagus nerve electrical stimulation during the surgery while the other half will get placebo therapy

ELIGIBILITY:
Inclusion Criteria:

* over 65 years old
* ability to communication
* hip or kneel replacement
* willing to participate in the study
* ASA I-II

Exclusion Criteria:

* with cerebral disorders or disease
* cognitive impairment before surgery
* with mental disease
* unable to communication
* severe eyes or ears impairment
* surgery performed in the past 30 days
* Bradycardia，II°AVB，III°AVB，severe heart, liver and kidney dysfunction
* severe skin disease
* refuse to enter the study

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of perioperative neurocognitive disorders | one month
  make different scale before and after operation to evaluate neurocognitive changes in experiment group and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Diansan Su, Shanghai, Shanghai Municipality, China